CLINICAL TRIAL: NCT02871869
Title: Cinobufacini Tablets Combined With R-CHOP Protocol (Rituximab + Vindesine + Cyclophosphamide + Epirubicin + Prednisone)/CHOP in Treatment of Diffuse Large B Cell Lymphoma: A Phase II Randomized, Controlled and Multi-center Study
Brief Title: Cinobufacini Tablets Combined With Chemotherapeutic Protocol in Treatment of Diffuse Large B Cell Lymphoma
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xinjiang Medical University (Other)
Responsible Party: Principal Investigator, Shun-E Yang, Xinjiang Medical University, Xinjiang Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XinjiangMU2016(015)V2.0
Record Dates: First submitted 2016-08-12; First posted 2016-08-18 (Estimated); Last update posted 2017-07-17 (Actual); Status verified 2017-07

CONDITIONS: Diffuse, Large B-Cell, Lymphoma
Keywords: Cinobufacini Tablets; CHOP protocol
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Vindesine; Cyclophosphamide; Epirubicin; Prednisone; huachansu; Buformin; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Control group A (Active Comparator): Control group A was treated with single R-CHOP protocol[Rituximab 375mg/㎡,one day before CHOP protocol, CHOP protocol included vindesine 3 mg/㎡ (maximum dosage: <4mg) d1 plus cyclophosphamide 750 mg/㎡ d1 plus Epirubicin 60 mg/㎡ d1 plus prednisone tablets 100 mg, d1～5], 21 d as a cycle, for 4～6 cycles.
  Interventions: Drug: vindesine; Drug: cyclophosphamide; Drug: Epirubicin; Drug: prednisone tablets; Drug: Rituximab
- Trial group A (Experimental): Trial group A was treated with Cinobufacini Tablets combined with R-CHOP protocol[Rituximab 375mg/㎡,one day before CHOP protocol, CHOP protocol included vindesine 3 mg/㎡ (maximum dosage: <4mg) d1 plus cyclophosphamide 750 mg/㎡ d1 plus Epirubicin 60 mg/㎡d1 plus prednisone tablets 100 mg, d1～5], 21 d as a cycle, for 4～6 cycles.
  Interventions: Drug: vindesine; Drug: cyclophosphamide; Drug: Epirubicin; Drug: prednisone tablets; Drug: Cinobufacini Tablets; Drug: Rituximab
- Control group B (Active Comparator): Control group B was treated with single CHOP protocol[vindesine 3 mg/㎡ (maximum dosage: <4mg) d1 plus cyclophosphamide 750 mg/㎡ d1 plus Epirubicin 60 mg/㎡ d1 plus prednisone tablets 100 mg, d1～5], 21 d as a cycle, for 4～6 cycles.
  Interventions: Drug: vindesine; Drug: cyclophosphamide; Drug: Epirubicin; Drug: prednisone tablets
- Trial group B (Experimental): Trial group B was treated with Cinobufacini Tablets combined with CHOP protocol[vindesine 3 mg/㎡ (maximum dosage: <4mg) d1 plus cyclophosphamide 750 mg/㎡ d1 plus Epirubicin 60 mg/㎡ d1 plus prednisone tablets 100 mg, d1～5], 21 d as a cycle, for 4～6 cycles.
  Interventions: Drug: vindesine; Drug: cyclophosphamide; Drug: Epirubicin; Drug: prednisone tablets; Drug: Cinobufacini Tablets

INTERVENTIONS:
Drug: vindesine — 3 mg/㎡ (maximum dosage: <4mg), d1, 21 d as a cycle, for 4～6 cycles
  Other Names: eldisine
Drug: cyclophosphamide — 750 mg/㎡, d1, 21 d as a cycle, for 4～6 cycles
  Other Names: endoxan
Drug: Epirubicin — 60 mg/㎡, d1, 21 d as a cycle, for 4～6 cycles
  Other Names: EPI
Drug: prednisone tablets — 100 mg, d1～5, 21 d as a cycle, for 4～6 cycles
  Other Names: metacortandracin
Drug: Cinobufacini Tablets — 0.3 g per tablet, 3 tablets per time, tid., p.o., until progressive disease or intolerable drug toxicities
  Other Names: buformin
  Arms: Trial group A; Trial group B
Drug: Rituximab — 375mg/㎡,one day before CHOP protocol
  Other Names: RTX
  Arms: Control group A; Trial group A

SUMMARY:
Diffuse large B cell lymphoma (DLBCL), as the most common subtype non-Hodgkin lymphoma (NHL), has great heterogeneity in clinical manifestations, histological morphology and prognosis. R-CHOP Protocol (Rituximab + Vindesine + Cyclophosphamide + Epirubicin + Prednisone) is the gold therapeutic criteria for patients with NHL, and it is also used as the first-line treatment for patients with DLBCL. After treatment, 50％～60％of patients with DLBCL receive complete remission (CR), 30％～40％ recurrent and 10% will never be cured due to initial and secondary drug tolerance. This study aimed to explore whether Cinobufacini Tablets had synergistic effect in the treatment of DLBCL, and whether its action was in close association with the positive expression of Na+/K+-ATPase α3, and to observe the rates of adverse reactions induced by Cinobufacini Tablets during treatment.

DETAILED DESCRIPTION:
Diffuse large B cell lymphoma (DLBCL), as the most common subtype non-Hodgkin lymphoma (NHL), accounts for 30％～40％ of adults with NHL, and has great heterogeneity in clinical manifestations, histological morphology and prognosis. R-CHOP Protocol (Rituximab + Vindesine + Cyclophosphamide + Epirubicin + Prednisone) is the gold therapeutic criteria for patients with NHL, and it is also used as the first-line treatment for patients with DLBCL. After treatment, 50％～60％of patients with DLBCL receive complete remission (CR), 30％～40％ recurrent and 10% will never be cured due to initial and secondary drug tolerance. The study of Tao Wu et al in domestic showed that cinobufacini combined with CHOP protocol had excellent efficacy in the treatment of NHL, with response rate reaching up to 91.7%, and the adverse reactions were mild and tolerable, whereas the response rate of single CHOP was only 62.5%. In the clinical practice of our studies, it was also found that some patients with recurrent DLBCL NHL also had shrunken or disappeared tumors and a survival time of more than 2 years after single administration of cinobufacini tablets for 3~6 months following the withdrawal of chemotherapy. This study aimed to explore whether Cinobufacini Tablets had synergistic effect in the treatment of DLBCL, and whether its action was in close association with the positive expression of Na+/K+-ATPase α3, and to observe the rates of adverse reactions induced by Cinobufacini Tablets during treatment.

ELIGIBILITY:
For control and trial groups A:

Inclusion Criteria:

* Patients aged 18-70 years old;
* Patients with eastern Collaborative Oncology Group (ECOG) performance status (PS) score: 0～3 points;
* International prognostic index (IPI): ≤3 points;
* Patients who were diagnosed as diffuse large B cell lymphoma (DLBCL) with initial treatment by histopathology;
* Patients with more than 1 measurable nidus (common CT or MRI scanning diameter ≥ 20 mm, and spiral CT scanning diameter ≥ 10 mm);
* Patients without dysfunction of important organs, and had normal blood routine, hepatorenal function and cardiac function. White blood cell count (WBC) ≥4.0×109/L, neutrophil count ≥1.5×109/L; platelet (PLT) count ≥100×109/L; hemoglobin (HGB) ≥95g/L; serum bilirubin (Bil) ≤1.5 folds of the upper limit of normal value, alanine transaminase (ALT) and aspartate aminotransferase (AST) ≤2 folds of the upper limit of normal value, and serum creatinine (Scr) ≤1.5mg/dl;
* Patients with expected survival time>3 months;
* Patients who were well informed of this study and signed the informed consent forms.
* Patients who received administration of Rituximab.

Exclusion Criteria:

* Patients who did not conform to above criteria;
* Patients who were receiving other anti-cancer therapies;
* Patients with DLBCL affected by primary breast gland, lung, testis, bone, peri-orbit, peri-spine, central nerve system and bone marrow;
* Patients with double expression, double strike, trinary expression and trinary strike and CD5+;
* Patients complicated with other non-DLBCL primary malignant tumors;
* Patients who had poor compliance with their families;
* Patients with one of the following conditions: uncontrolled metastatic nidi of central nerve system, dysfunction of important organs and severe cardiac diseases like congestive heart failure, uncontrollable arrhythmia, angina pectoris that needed long-term drug administration, valvular heart diseases, myocardial infarction and refractory hypertension, pregnancy or lactation, chronic infectious wounds, and history of uncontrollable psychological diseases.
* Patients had previous history of treatment with Cinobufacini Tablets.

For control and trial groups B

Inclusion Criteria:

* Patients aged 18-70 years old;
* Patients with eastern Collaborative Oncology Group (ECOG) performance status (PS) score: 0～3 points;
* International prognostic index (IPI): ≤3 points;
* Patients who were diagnosed as diffuse large B cell lymphoma (DLBCL) with initial treatment by histopathology;
* Patients with more than 1 measurable nidus (common CT or MRI scanning diameter ≥ 20 mm, and spiral CT scanning diameter ≥ 10 mm);
* Patients without dysfunction of important organs, and had normal blood routine, hepatorenal function and cardiac function. White blood cell count (WBC) ≥4.0×109/L, neutrophil count ≥1.5×109/L; platelet (PLT) count ≥100×109/L; hemoglobin (HGB) ≥95g/L; serum bilirubin (Bil) ≤1.5 folds of the upper limit of normal value, alanine transaminase (ALT) and aspartate aminotransferase (AST) ≤2 folds of the upper limit of normal value, and serum creatinine (Scr) ≤1.5mg/dl;
* Patients with expected survival time>3 months;
* Patients who were well informed of this study and signed the informed consent forms.
* Patients who did not receive administration of Rituximab.

Exclusion Criteria:

* Patients who did not conform to above criteria;
* Patients who were receiving other anti-cancer therapies;
* Patients with DLBCL affected by primary breast gland, lung, testis, bone, peri-orbit, peri-spine, central nerve system and bone marrow;
* Patients with double expression, double strike, trinary expression and trinary strike and CD5+;
* Patients complicated with other non-DLBCL primary malignant tumors;
* Patients who had poor compliance with their families;
* Patients with one of the following conditions: uncontrolled metastatic nidi of central nerve system, dysfunction of important organs and severe cardiac diseases like congestive heart failure, uncontrollable arrhythmia, angina pectoris that needed long-term drug administration, valvular heart diseases, myocardial infarction and refractory hypertension, pregnancy or lactation, chronic infectious wounds, and history of uncontrollable psychological diseases.
* Patients had previous history of treatment with Cinobufacini Tablets.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 316 (Estimated)
Dates: Start 2016-09; Primary Completion 2018-09 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | 3 years
  3-year Progression-free survival (PFS) defined as the ratio of study subjects who had disease progression or died within 3 years from the start of randomization.

SECONDARY OUTCOMES:
Overall response rate (ORR) | 2 years
  Overall response rate (ORR) that defined as the total ratio of study subjects with complete response, complete response unconfirmed and partial response after treatment. ORR=(CR+ CRu+ PR)cases/total cases×100%.
overall survival rate (OS) | 3 years
  3-year overall survival rate (OS) that defined as the ratio of study subjects who survived 3 years after randomization
Safety and Tolerability | 2 years
  Incidence of Treatment-Emergent adverse events
Relationship between synergistic effect of Cinobufacini Tablets and expression of Na+/K+-ATPase α3 | 2 years
  Relationship between synergistic effect of Cinobufacini Tablets and expression of Na+/K+-ATPase α3

CONTACTS AND LOCATIONS:
Overall Officials: Shun-E Yang, Professor, Study Chair — Cancer Hospital Affiliated to Xinjiang Medical University
Locations (1):
- Cancer Hospital Affiliated to Xinjiang Medical University, Ürümqi, Xinjiang, China

IPD SHARING:
Plan to Share IPD: No